CLINICAL TRIAL: NCT07304479
Title: Effects of Sevoflurane Versus Desflurane Anesthesia Under Protective Mechanical Ventilation for Robotic Assisted Surgery on Airway Plateau Pressure: a Randomized, Prospective, Blinded Pilot Study
Brief Title: Effects of Sevoflurane Versus Desflurane Anesthesia Under Protective Mechanical Ventilation for Robotic Assisted Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Aliki Tympa, Assistant Professor of Anesthesiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 705/25-07-2025
Record Dates: First submitted 2025-09-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Mechanics; Intraoperative
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Volatile Anesthetic) (Active Comparator)
  Interventions: Drug: Sevoflurane (Volatile Anesthetic)
- Deslfurane (Volatile Anesthetic) (Active Comparator)
  Interventions: Drug: Desflurane (volatile anesthetic)

INTERVENTIONS:
Drug: Sevoflurane (Volatile Anesthetic) — Sevoflurane for robotic assisted laparoscopic surgery
  Arms: Sevoflurane (Volatile Anesthetic)
Drug: Desflurane (volatile anesthetic) — Desflurane for robotic assisted laparoscopic surgery
  Arms: Deslfurane (Volatile Anesthetic)

SUMMARY:
Inhalational anesthetics, when used in abdominal surgery, offer advantages of lung protection and reduced alveolar inflammation. There is little literature, however, in the comparative use of sevoflurane versus desflurane anesthesia in patients undergoing abdominal robotic-assisted surgery and their effects on lung mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 87 years
* Undergoing elective robotic-assisted abdominal surgery
* ASA physical status I-III

Exclusion Criteria:

* ASA IV or V
* Emergency surgery
* Renal insufficiency
* Clinically significant respiratory disease
* Cardiomyopathy
* Uncontrolled hypertension

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
airway plateau pressure | Perioperatively
  Airway plateau pressure (cmH2O) as displayed on the anesthesia ventilator at the specified time points will be recorded for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini Melemeni, Professor, Study Director — Aretaieion University Hospital, National And Kapodistrian University Of Athens
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herling SF, Dreijer B, Wrist Lam G, Thomsen T, Moller AM. Total intravenous anaesthesia versus inhalational anaesthesia for adults undergoing transabdominal robotic assisted laparoscopic surgery. Cochrane Database Syst Rev. 2017 Apr 4;4(4):CD011387. doi: 10.1002/14651858.CD011387.pub2. PMID 28374886